CLINICAL TRIAL: NCT00623480
Title: Randomized, Controlled, Parallel, Prospective Trial to Evaluate the Effect of Secondary Prophylaxis With rFVIII Therapy in Severe Hemophilia A Adult and/or Adolescent Subjects, as Applicable, Compared to That of Episodic Treatment
Brief Title: Trial to Evaluate the Effect of Secondary Prophylaxis With rFVIII Therapy in Severe Hemophilia A Adult and/or Adolescent Subjects Compared to That of Episodic Treatment
Acronym: SPINART
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Bayer (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 12800; 2008-000985-21 (EudraCT Number)
Record Dates: First submitted 2008-02-04; First posted 2008-02-26 (Estimated); Results first posted 2013-08-07 (Estimated); Last update posted 2014-11-17 (Estimated); Status verified 2014-11

CONDITIONS: Hemophilia A
Keywords: Hemophilia A
MeSH Terms: conditions — Hemophilia A | interventions — Factor VIII; F8 protein, human; BAY 14-2222

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Recombinant Factor VIII prophylaxis treatment (Experimental): Participants received 25 IU/kg of Recombinant Factor VIII (Kogenate FS, BAY14-2222) intravenously (IV), 3 times per week. Dose escalation steps by 5 IU/kg (to 30 IU/kg or 35 IU/kg maximum) for patients exhibiting a bleeding frequency of 12 bleeding episodes per year or greater.
  Interventions: Biological: Recombinant Factor VIII (Kogenate FS, BAY14-2222)
- Recombinant Factor VIII on-demand treatment (Experimental): Participants received Recombinant Factor VIII (Kogenate FS, BAY14-2222) IV for bleeds in accordance with package insert instructions and study physician recommendations.
  Interventions: Biological: Recombinant Factor VIII (Kogenate FS, BAY14-2222)

INTERVENTIONS:
Biological: Recombinant Factor VIII (Kogenate FS, BAY14-2222) — Prophylaxis treatment includes three times per week administration of 25 IU/kg of Kogenate FS. Dose escalation steps by 5 IU/kg (to 30 IU/kg or 35 IU/kg maximum) exhibiting a bleeding frequency of 12 bleeding episodes per year or greater.
  Arms: Recombinant Factor VIII prophylaxis treatment
Biological: Recombinant Factor VIII (Kogenate FS, BAY14-2222) — Treated according to the Kogenate FS package insert indications and study physician recommendations
  Arms: Recombinant Factor VIII on-demand treatment

SUMMARY:
To evaluate the effect of secondary prophylaxis as compared to episodic treatment on bleeding frequency (number of bleeds per year) and on joint damage.

ELIGIBILITY:
Inclusion Criteria:

* Males aged 12 to 50 years (US and Argentina)
* Males aged 18 to 50 years (other countries)
* Subjects with severe hemophilia A (<1% FVIII:C) as confirmed by the central lab from a sample obtained at least 96 hours after FVIII administration wash-out. Allow for the inclusion of a maximum of 10% (n=8) of patients with 1-2% FVIII:C baseline levels as long as they exhibit clinical severity and comply with all other inclusion criteria.
* Subjects with at least 150 prior exposure days with any FVIII
* Subjects who have been on episodic treatment and no known regular prophylaxis treatment for more than 12 consecutive months in the previous 5 years
* Subjects with 6 to 24 bleeding events and/or treatments in the previous 6 months prior to study entry which are documented and available in the subjects medical records. Documentation can include records from previous physicians, specific home treatment records, emergency room or hospital records, x-ray reports, etc. The investigator can also document with a detailed note the number of bleeds reported by the subject in the last 6 months.
* Subjects with inhibitor formation surveillance (inhibitor or recovery testing) over the ten years prior to enrollment documented by the investigator and who do not have a history of any of the following:

  * A positive inhibitor titer of 5.0 Bethesda Unit (BU) or greater by either BU assay system at any time since first exposure to exogenous factor VIII
  * A positive inhibitor test result of 1.0 or greater performed by the original BU assay at any time in the past 10 years (A subject can have more than one positive inhibitor test of 0.6 or greater by the original BU assay test but all must be less than 1.0 BU using the original BU assay.)
  * A positive inhibitor test result of 0.6 or greater performed by the Nijmegen method at any time in the past 10 years
* Subjects with no inhibitor activity by Nijmegen-modified Bethesda assay, either positive (> 0.6 BU is considered positive) or borderline (> 0.3 and < 0.6 BU is considered borderline) as measured in the current study reference laboratory

Exclusion Criteria:

* Subjects with any other bleeding disease besides hemophilia A (i.e. von Willebrand disease)
* Subjects with thrombocytopenia (platelets < 100,000/mm3)
* Subjects with abnormal renal function (Cockcroft-Gault Creatinine Clearance value of 60 mL/min or lower)
* Subjects with active hepatic disease (Aspartate aminotransferase [AST] or Alanine aminotransferase [ALT] > 5xUpper Limit of Normal (ULN))
* Subjects on treatment with immunomodulatory agents within the last 3 months prior to study entry or during the study (the following drugs are however allowed: interferon-a treatment for Hepatitis C virus (HCV), Highly active anti-retroviral therapy (HAART) therapy for human immunodeficiency virus (HIV) and/or a total of two courses of pulse treatment with steroids for a maximum of 7 days at 1mg/kg or less)
* Subjects with an absolute CD4 lymphocyte cell count < 200 cells/mm3 (due to HIV, HCV or another suspected medical condition)
* Subjects with known hypersensitivity to rFVIII, mouse or hamster proteins
* Subjects who are receiving or had received other experimental drugs within 1 month prior to study entry
* Subjects who require any pre-medication to tolerate FVIII injections (e.g. anti-histamines)
* Subjects who are unwilling to comply with study visits or either of the possible treatment regimens
* Subjects who have a planned orthopedic intervention to be performed during the study that may substantially affect bleeding (e.g. surgical or chemical or radiological synovectomy)
* Subjects who are not suitable for participation in this study for any reason, according to the Investigator
* Subjects who have poor joint status as defined by routine need for a wheelchair or unable to ambulate without the assistance of a brace, cane or crutches
* Three or more joints that are already fused or "frozen" also called ankylosis

Ages: 12 Years to 50 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 84 (Actual)
Dates: Start 2008-03; Primary Completion 2011-09 (Actual); Study Completion 2013-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Bayer Study Director, Study Director — Bayer
Locations (35):
- United States (26):
  - Tucson, Arizona
  - Little Rock, Arkansas
  - Orange, California
  - Sacramento, California
  - Aurora, Colorado
  - Washington D.C., District of Columbia
  - Orlando, Florida
  - Atlanta, Georgia
  - Chicago, Illinois
  - Indianapolis, Indiana
  - Iowa City, Iowa
  - Louisville, Kentucky
  - Boston, Massachusetts
  - Detroit, Michigan
  - Minneapolis, Minnesota
  - Kansas City, Missouri
  - Las Vegas, Nevada
  - Newark, New Jersey
  - New York, New York
  - Cleveland, Ohio
  - Hershey, Pennsylvania
  - Pittsburgh, Pennsylvania
  - Knoxville, Tennessee
  - Houston, Texas
  - Salt Lake City, Utah
  - Milwaukee, Wisconsin
- Argentina (2):
  - Buenos Aires, Ciudad Auton. de Buenos Aires
  - Rosario, Santa Fe Province
- Bulgaria (3):
  - Plovdiv
  - Sofia
  - Varna
- Romania (4):
  - Timișoara, Timiș County
  - Brasov
  - Bucharest
  - Constanța

REFERENCES:
- [Result] Manco-Johnson MJ, Kempton CL, Reding MT, Lissitchkov T, Goranov S, Gercheva L, Rusen L, Ghinea M, Uscatescu V, Rescia V, Hong W. Randomized, controlled, parallel-group trial of routine prophylaxis vs. on-demand treatment with sucrose-formulated recombinant factor VIII in adults with severe hemophilia A (SPINART). J Thromb Haemost. 2013 Jun;11(6):1119-27. doi: 10.1111/jth.12202. PMID 23528101
- [Derived] Manco-Johnson MJ, Lundin B, Funk S, Peterfy C, Raunig D, Werk M, Kempton CL, Reding MT, Goranov S, Gercheva L, Rusen L, Uscatescu V, Pierdominici M, Engelen S, Pocoski J, Walker D, Hong W. Effect of late prophylaxis in hemophilia on joint status: a randomized trial. J Thromb Haemost. 2017 Nov;15(11):2115-2124. doi: 10.1111/jth.13811. Epub 2017 Oct 10. PMID 28836341

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Recombinant Factor VIII Prophylaxis Treatment | Recombinant Factor VIII On-demand Treatment
Started | 42 | 42
Completed | 35 | 35
Not Completed | 7 | 7
Not completed — Lost to Follow-up | 0 | 1
Not completed — Withdrawal by Subject | 2 | 4
Not completed — Lack of Efficacy | 1 | 0
Not completed — Non-compliant with study medication | 4 | 0
Not completed — Protocol Violation | 0 | 1
Not completed — Site closed by sponsor | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Recombinant Factor VIII Prophylaxis Treatment | Recombinant Factor VIII On-demand Treatment | Total
Number analyzed (Participants) | 42 | 42 | 84
Age, Continuous [Mean (Standard Deviation); unit: Years] | 30.6 (8.8) | 30.7 (9.7) | 30.6 (9.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0
  Male | 42 | 42 | 84
Number of bleeds during last 6 months [Mean (Standard Deviation); unit: Bleeds] | 10.0 (4.4) | 12.2 (5.1) | 11.1 (4.8)
Number of patients with target joints, Yes/No [Number; unit: Participants] — A 'target joint' is a particular joint that has experienced repeated bleeds or at least four bleeds into one joint within a six month period.
  Participants
    Yes | 28 | 31 | 59
    No | 14 | 11 | 25

OUTCOME MEASURES:

1. Primary Outcome: Bleeding Frequency (Number of Total Bleeds)
Time Frame: After the last enrolled patient has been in the study for 1 year. At the cut-off, the median follow-up duration was 616 days (minimum was 111 days and maximum was 1109 days)
Population: ITT (Intent-to-treat) Population
Measure: Median (Full Range); unit: Bleeds
Arm/Group | Recombinant Factor VIII Prophylaxis Treatment | Recombinant Factor VIII On-demand Treatment
Number analyzed (Participants) | 42 | 42
Bleeds | 0 [0 to 57] | 54.5 [0 to 149]
Statistical Analysis 1: Comparison: Recombinant Factor VIII Prophylaxis Treatment vs Recombinant Factor VIII On-demand Treatment; Test type: Superiority or Other; p < 0.0001, Negative Binomial Regression Model; Adjusted for time of follow-up; Ratio (On-Demand vs. Prophylaxis) = 14.7, 95% CI 2-sided [8.1 to 26.5]

2. Secondary Outcome: Change From Baseline to 3 Years in the MRI (Magnetic Resonance Imaging) Scale.
Description: The Extended MRI Scale total score has a range between 0 (normal unaffected joint) to 45 (maximal joint damage) points. It is composed of 2 domains, the soft tissue domain with a maximum of 9 points and the osteochondral domain with a maximum of 36 points. A single score for each subject was to be calculated from the sum of both domains and the average over all joints for the Extended MRI endpoint. Higher MRI score denotes greater joint structure damage thus a positive change from baseline means worsening.
Time Frame: Baseline and 3 years
Population: Full Analysis Set
Measure: Least Squares Mean (95% Confidence Interval); unit: Scores on a scale
Arm/Group | Recombinant Factor VIII Prophylaxis Treatment | Recombinant Factor VIII On-demand Treatment
Number analyzed (Participants) | 41 | 38
Scores on a scale | 0.79 [0.27 to 1.32] | 0.96 [0.34 to 1.58]
Statistical Analysis 1: Comparison: Recombinant Factor VIII Prophylaxis Treatment vs Recombinant Factor VIII On-demand Treatment; Test type: Superiority or Other; p = 0.6614, Based on cLDA model; Adjusted for presence/absence of target joint and prior 6 month bleeding frequency; estimated diff (prohylaxis vs. OD) = -0.17, 95% CI 2-sided [-0.92 to 0.59]

3. Secondary Outcome: Change From Baseline to 3 Years in the Colorado Adult Joint Assessment Scale
Description: The total joint score is derived for each of six joints: left and right sides for knees (score: 0-25), ankles (score: 0-25), and elbows (score: 0-21). Higher CAJAS (Colorado Adult Joint Assessment Scale) score denotes greater joint structure damage thus a positive change from baseline means worsening. CAJAS total score is the sum of all 6 joints, ranging from 0 (best possible outcome) to 142 (worst possible outcome).
Time Frame: Baseline and 3 years
Population: Full Analysis Set
Measure: Least Squares Mean (95% Confidence Interval); unit: Scores on a scale
Arm/Group | Recombinant Factor VIII Prophylaxis Treatment | Recombinant Factor VIII On-demand Treatment
Number analyzed (Participants) | 42 | 42
Scores on a scale | -0.31 [-0.79 to 0.18] | 0.63 [0.08 to 1.18]
Statistical Analysis 1: Comparison: Recombinant Factor VIII Prophylaxis Treatment vs Recombinant Factor VIII On-demand Treatment; Test type: Superiority or Other; p = 0.0072, Based on cLDA model; Adjusted for presence/absence of target joint and prior 6 month bleeding frequency; estimated diff (prohylaxis vs. OD) = -0.94, 95% CI 2-sided [-1.61 to -0.26]

4. Other Pre Specified Outcome: Change From Baseline to 3 Years in the Physical Functioning Domain of the Haemo-QoL-A
Description: The Haemo-QoL-A total score as well as each of its domains have a range between 0 (worst Quality of Life) and 100 (best Quality of Life) points. Therefore, a higher Haemo-QoL-A score denotes greater Quality of Life.
Time Frame: Baseline and 3 years
Population: Full Analysis Set
Measure: Least Squares Mean (95% Confidence Interval); unit: Scores on a scale
Arm/Group | Recombinant Factor VIII Prophylaxis Treatment | Recombinant Factor VIII On-demand Treatment
Number analyzed (Participants) | 41 | 42
Scores on a scale | 7.86 [1.79 to 13.92] | -5.30 [-11.97 to 1.37]
Statistical Analysis 1: Comparison: Recombinant Factor VIII Prophylaxis Treatment vs Recombinant Factor VIII On-demand Treatment; Test type: Superiority or Other; Based on cLDA model — no p-values computed; Adjusted for presence/absence of target joint and prior 6 month bleeding frequency; estimated diff (prohylaxis vs. OD) = 13.15, 95% CI 2-sided [5.23 to 21.08]

ADVERSE EVENTS:
Time Frame: From randomization until Month 37.
Arm/Group | Recombinant Factor VIII Prophylaxis Treatment | Recombinant Factor VIII On-demand Treatment
Serious Adverse Events (participants affected / at risk) | 9/42 | 11/42
Other Adverse Events (participants affected / at risk) | 11/42 | 28/42
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Recombinant Factor VIII Prophylaxis Treatment (N=42) | Recombinant Factor VIII On-demand Treatment (N=42)
Anaemia (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Phimosis (Congenital, familial and genetic disorders) | 0 (0) | 1 (1)
Peritoneal haemorrhage (Gastrointestinal disorders) | 1 (1) | 0 (0)
Retroperitoneal haematoma (Gastrointestinal disorders) | 1 (1) | 0 (0)
Tooth impacted (Gastrointestinal disorders) | 1 (1) | 0 (0)
Appendicitis (Infections and infestations) | 2 (2) | 1 (1)
Device related infection (Infections and infestations) | 1 (1) | 0 (0)
Peritonsillar abscess (Infections and infestations) | 1 (1) | 0 (0)
Pilonidal cyst (Infections and infestations) | 1 (1) | 0 (0)
Fibula fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Humerus fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Meniscus injury (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Stab wound (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Tibia fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Dehydration (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Haemarthrosis (Musculoskeletal and connective tissue disorders) | 0 (0) | 2 (2)
Joint contracture (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Joint lock (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Joint range of motion decreased (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Muscle haemorrhage (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Migraine (Nervous system disorders) | 1 (1) | 0 (0)
Suicidal ideation (Psychiatric disorders) | 1 (1) | 0 (0)
Balanitis (Reproductive system and breast disorders) | 0 (0) | 1 (1)
Haematoma (Vascular disorders) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Recombinant Factor VIII Prophylaxis Treatment (N=42) | Recombinant Factor VIII On-demand Treatment (N=42)
Dental caries (Gastrointestinal disorders) | 0 (0) | 3 (3)
Dyspepsia (Gastrointestinal disorders) | 0 (0) | 3 (3)
Toothache (Gastrointestinal disorders) | 3 (3) | 2 (3)
Pyrexia (General disorders) | 1 (2) | 5 (6)
Influenza (Infections and infestations) | 2 (2) | 7 (7)
Nasopharyngitis (Infections and infestations) | 2 (2) | 7 (8)
Pharyngitis (Infections and infestations) | 0 (0) | 3 (4)
Upper respiratory tract infection (Infections and infestations) | 1 (1) | 3 (5)
Vitamin D deficiency (Metabolism and nutrition disorders) | 0 (0) | 3 (3)
Arthralgia (Musculoskeletal and connective tissue disorders) | 5 (7) | 5 (6)
Back pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 4 (5)
Myalgia (Musculoskeletal and connective tissue disorders) | 3 (3) | 1 (1)
Headache (Nervous system disorders) | 2 (2) | 7 (12)
Cough (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 3 (3)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 3 (3)
Hypertension (Vascular disorders) | 0 (0) | 3 (3)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Investigator must send a draft manuscript of the publication or abstract to the Sponsor sixty days in advance of submission in order to obtain written approval prior to submission of the final version for publication. In case of a difference of opinion between the Sponsor and the Investigator(s), the contents of the publication will be discussed in order to find a solution which satisfies both parties.